CLINICAL TRIAL: NCT07171996
Title: Research on the Optimization of Treatment for Spinal Metastases With Radioactive Particle Implantation Using TPS and Mechanical Dual Simulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960HP20250410
Record Dates: First submitted 2025-09-11; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Bone Metastases in Subjects With Advanced Cancer
Keywords: tps; dynamics; osseous metastasis

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, open-label trial comparing dual-simulation planning (TPS + patient-specific biomechanical FE model) versus conventional TPS for image-guided radioactive seed implantation in bone metastases.
Masking Description: Masking: None (Open Label). Due to the procedural nature of seed implantation, participants and treating clinicians cannot be blinded. To reduce bias, key outcomes are assessed under blinded procedures: (1) centralized, de-identified imaging and dosimetry review by independent radiologists/physicists blinded to allocation; (2) pain and QoL collected via standardized instruments by staff not involved in planning, with pre-specified analgesic adjustment rules; (3) an independent endpoint adjudication committee and the statistical analysis team remain blinded to group assignment, using Arm A/B codes. Allocation is concealed until plan finalization; intraoperative teams are unblinded. Participants are instructed not to disclose perceived assignment to assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - TPS + Biomechanical Dual-Simulation (Experimental): Single-group assignment using the dual-simulation planning workflow integrating TPS with patient-specific finite element modeling to optimize dose distribution and mechanical safety (fracture risk, needle stability, seed migration). Image-guided implantation is performed per optimized plan; postoperative CT provides dosimetric verification. Outcomes include pain response, dosimetry, biomechanics-related events, and safety.
  Interventions: Other: Dual-Simulation TPS + Biomechanical Planning
- Active Comparator - Conventional TPS (Active Comparator): Preoperative planning using conventional TPS per institutional standards to meet dosimetric goals and OAR constraints; no biomechanical modeling. Image-guided implantation per plan; postoperative CT for seed localization and dosimetric verification. Follow-up schedule identical to the
  Interventions: Other: Conventional TPS Planning

INTERVENTIONS:
Other: Dual-Simulation TPS + Biomechanical Planning — Combines TG-43-based TPS with a patient-specific FE biomechanical model to optimize needle paths and seed placement considering OAR limits, fracture risk, needle stability, and seed migration risk.
  Arms: Experimental - TPS + Biomechanical Dual-Simulation
Other: Conventional TPS Planning — Conventional TPS-driven plan per institutional practice; no biomechanical modeling.
  Arms: Active Comparator - Conventional TPS

SUMMARY:
This prospective, open-label randomized trial evaluates a dual-simulation planning strategy that combines standard brachytherapy TPS with patient-specific biomechanical modeling for radioactive seed implantation in bone metastases. The approach aims to improve dose coverage while accounting for fracture risk, needle path stability, and seed migration. Eligible patients with painful and/or progressive bone metastases are randomized to dual-simulation planning versus conventional TPS. All undergo image-guided implantation with post-implant dosimetric verification and standardized follow-up. The primary endpoint is 3-month pain response (BPI/VAS, adjusted for analgesic use). Secondary endpoints include dosimetry (D90, V100, CI, HI), local control/progression, seed migration, skeletal-related events and fractures, SINS and functional status, quality of life, procedure-related complications (CTCAE v5.0), and procedure metrics. We hypothesize the dual-simulation strategy will enhance dosimetric quality and reduce biomechanics-related complications, improving pain and function.

DETAILED DESCRIPTION:
This study aims to evaluate a "dual-simulation" optimization strategy that combines a brachytherapy treatment planning system (TPS) with biomechanical modeling to improve the feasibility, safety, and effectiveness of radioactive seed implantation for bone metastases (palliative/local control). Conventional TPS is primarily dose-centric and may not adequately account for the mechanical stability of metastatic bone lesions, feasibility of needle trajectories, or risk of seed migration, potentially leading to suboptimal dose distribution or increased post-procedural biomechanics-related adverse events. To address this gap, we integrate a patient-specific finite element biomechanical model into standard TPS to predict load-bearing behavior, fracture risk, needle path stability, and seed migration risk, enabling iterative, dose-mechanics constrained plan optimization.

This is a prospective, open-label, randomized controlled trial comparing "TPS + biomechanical dual-simulation" versus conventional TPS. Eligible participants are patients with bone metastases who meet indications for radioactive seed implantation and have pain and/or risk of local progression. In the experimental arm, preoperative imaging segmentation and individualized biomechanical modeling inform coupled optimization of needle trajectories and seed distributions; the control arm receives standard TPS-based planning. All patients undergo image-guided implantation, with post-implant dosimetric verification and standardized follow-up.

The primary endpoint is pain response at 3 months (per BPI or VAS, accounting for changes in analgesic use). Secondary endpoints include dosimetric parameters (e.g., D90, V100, conformity index [CI], homogeneity index [HI]), local control rate and time to progression, seed migration incidence, skeletal-related events (SREs) and pathologic fracture incidence/time, changes in SINS score and functional status (e.g., ECOG, TESS), quality of life (EORTC QLQ-C30), procedure-related complications (CTCAE v5.0), and procedure time/number of needle adjustments. Safety will be assessed at prespecified time points. Imaging will be performed at baseline, post-procedure, and during follow-up, with standardized post-implant dosimetric verification.

We hypothesize that the dual-simulation strategy will maintain or improve dose coverage and conformity while reducing seed migration and biomechanics-related complications, thereby improving pain relief and functional outcomes, and providing a more comprehensive, individualized optimization pathway for radioactive seed implantation in bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.

Radiologically or histologically confirmed bone metastasis with a lesion suitable for percutaneous radioactive seed implantation (e.g., I-125), per multidisciplinary assessment.

Indication for local palliation/control: moderate-to-severe pain at lesion (e.g., BPI/VAS ≥4) and/or imaging evidence of progression or high-risk features warranting local therapy.

Measurable/evaluable target lesion on CT/MRI; target location accessible for needle placement per institutional practice.

ECOG performance status 0-2.

Estimated life expectancy ≥3 months.

Adequate hemostasis: platelets ≥80×10^9/L, INR ≤1.5 (or per protocol), and able to hold/bridge anticoagulation as clinically indicated.

Adequate organ function to undergo the procedure and anesthesia/sedation per site standards.

Able to undergo required imaging (CT; MRI if applicable).

Willing and able to provide written informed consent and comply with follow-up.

For women of childbearing potential and men with partners of childbearing potential: agreement to use effective contraception during and for the protocol-defined period after implantation.

Exclusion Criteria:

* Need for urgent surgical decompression or stabilization (e.g., acute/impending neurologic compromise, unstable pathologic fracture) that precludes percutaneous implantation at this time.

Uncorrected coagulopathy or ongoing antithrombotic therapy that cannot be safely managed periprocedurally.

Active systemic or local infection at/near the planned access route.

Diffuse marrow replacement or extensive cortical destruction where percutaneous implantation is unsafe or unlikely to achieve local control without stabilization, per MDT judgment.

Prior radiation or surgery to the index lesion that, in the investigator's opinion, makes additional seed implantation unsafe or non-beneficial; postoperative bed without a discrete target for seed placement.

Known hypersensitivity to materials/agents required for the procedure (e.g., contrast) not amenable to premedication or alternative imaging.

Uncontrolled medical conditions posing prohibitive procedural risk (e.g., severe cardiopulmonary disease, uncontrolled hypertension/arrhythmia).

Pregnant or breastfeeding.

Inability to lie still or contraindications to required imaging/sedation not correctable.

Concurrent participation in another interventional study that could confound efficacy/safety assessment at the treated site.

Any condition that, in the investigator's judgment, would interfere with protocol adherence, safety monitoring, or outcome assessment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Response at 3 Months | Baseline (≤14 days pre-implant) and 3 months post-implant (±14 days)
  Proportion of participants achieving pain response at the treated site 3 months post-implant, defined as ≥2-point absolute reduction or ≥30% relative reduction from baseline in worst pain (BPI-SF item 3 or 0-10 VAS), without an increase in analgesic consumption; if analgesic use changes, response is adjudicated using standardized analgesic-adjusted criteria (e.g., IMMPACT-consistent rules with oral morphine equivalent dose). Pain is collected by trained staff blinded to allocation; centralized, de-identified adjudication applies. Primary analysis compares proportions between arms (risk difference and 95% CI; two-sided α=0.05). Time Frame: Baseline and 3 months post-implant.
Local Tumor Control (Treated Site) | 6 months (±30 days), 12 months (±45 days); exploratory at 24 months (±60 days)
  Proportion of participants without local progression at the treated lesion, assessed by centralized imaging review. Local progression is defined as any of: (a) ≥20% increase in maximal diameter or volumetric expansion on CT/MRI with an absolute increase of ≥5 mm; (b) new nodular enhancement or soft-tissue extension contiguous with the treated site; (c) unequivocal progression by MD Anderson bone response criteria; or (d) metabolic progression on PET-CT per PERCIST when available. Death without prior local progression is counted as failure in sensitivity analyses; primary analysis censors at last evaluable imaging. Results reported as local control rate and Kaplan-Meier estimates of time to local progression with 95% CIs. Imaging is reviewed by blinded independent radiologists/physicists

CONTACTS AND LOCATIONS:
Overall Officials: min 李 li, Study Director
Locations (1):
- The 960 Hospital of the People's Liberation Army of China, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data including baseline demographics and clinical characteristics; lesion site and imaging features; planning inputs (e.g., TPS parameters, seed model), dosimetry metrics (D90, V100, CI, HI), biomechanical model outputs (stress/strain maps summarized, fracture/migration risk scores), procedure details (needle count/paths, procedure time, intraoperative deviations), safety data (AEs/SAEs per CTCAE v5.0), analgesic use, pain scores (BPI/VAS), functional status (ECOG/TESS), quality of life (EORTC QLQ-C30), and imaging-derived efficacy endpoints (local control/progression dates and assessments). Dates will be shifted or bucketed to protect privacy; direct identifiers will be removed.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting documents will be available starting 12 months after the primary completion date or upon publication of the primary results, whichever occurs first, and will remain available for 5 years thereafter (extensions considered upon justified request).
Access Criteria: Qualified researchers with a methodologically sound proposal may request access. Required materials include a brief proposal and analysis plan, IRB/ethics approval or exemption (as applicable), and a signed Data Use Agreement. Requests are reviewed by the study's Data Access Committee within ~30 calendar days. Approved users will access a de-identified, analysis-ready dataset via a controlled-access secure environment; raw downloads are restricted. Available materials include: de-identified participant-level dataset, data dictionary/codebook, de-identification schema, redacted protocol, statistical analysis plan, blank CRFs, and analytic code used for primary endpoints (R/Python). Submit requests via the study data portal or email the IPD contact.